CLINICAL TRIAL: NCT01338389
Title: Influence of Oral Treatment With Citicoline for the Prevention of Radiation Optic Neuropathy in Patients Treated for Uveal Melanomas With Proton Beam Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Collaborators: DENSMORE pharmaceuticals (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 11-PP-04
Record Dates: First submitted 2011-04-18; First posted 2011-04-19 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2024-04

CONDITIONS: Uveal Melanoma
MeSH Terms: conditions — Uveal Melanoma | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CITICOLINE (Experimental): Daily oral administration of 800 mg citicoline
  Interventions: Dietary Supplement: CITICOLINE
- Placebo (Placebo Comparator): Daily oral administration of placebo
  Interventions: Dietary Supplement: PLACEBO

INTERVENTIONS:
Dietary Supplement: CITICOLINE — Oral administration of CITICOLINE:
  Form: Powder for solution Dosage: 800mg per day duration: 5 years
  Arms: CITICOLINE
Dietary Supplement: PLACEBO — Oral administration of placebo:
  Form: Powder for solution duration: 5 years
  Arms: Placebo

SUMMARY:
Proton beam irradiation is the treatment of choice for uveal melanomas. It has favorable results in causing tumor regression while preserving the eye. Optic neuropathy has emerged consistently as an irreversible cause of visual loss in proton beam irradiated eyes. No neuroprotective strategies are available at present.

Citicoline is a choline agent precursor available as a dietary supplement. Citicoline conferred acute neuroprotection and enhanced neuroplasticity in experimental stroke models. In ophthalmology, citicoline has demonstrated a significant action in improving retinal and cortical responses in patients with optic nerve diseases (glaucoma, ischemic optic neuropathy). Citicoline also exhibits a very low toxicity profile in humans.

The purpose of the study is to demonstrate whether daily oral administration of citicoline in patients treated for uveal melanomas with proton beam therapy, prevents or delays the occurrence of radiation optic neuropathy. Changes in visual acuity, Pattern ERG and visual evoked potentials are measured. The tolerability/safety of the product is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* uveal melanoma with posterior marge located at less than 3 mm of optic papilla
* uveal melanoma treated with proton beam therapy with irradiation of optic head nerve
* visual acuity before proton beam therapy over 30 letters (with ETDRS test)

Exclusion Criteria:

* antecedent of acute glaucoma with angle enclosure
* antecedent of chronical glaucoma with angle aperture
* antecedent of optic neuropathy optique of congenital, ischemic, inflammatory or other origins
* antecedent of neovascular glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-06-25 (Actual); Primary Completion 2017-06-29 (Actual); Study Completion 2017-06-29 (Actual)

PRIMARY OUTCOMES:
Occurrence and delay of occurrence of radiation optic neuropathy | Every 6 months
  Occurrence and delay of occurrence of radiation optic neuropathy in patients treated for uveal melanomas with proton beam therapy

SECONDARY OUTCOMES:
Visual function assessment | Every 6 months
  Best corrected visual acuity (ETDRS) ; Pattern ERG ; Visual Evoked potentials; adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie BAILLIF-GOSTOLI, MD, Principal Investigator — Ophtalmology department, Nice University Hospital
Locations (2):
- France (2):
  - CHU de NICE, Nice
  - Ophtalmology Departement, St Roch Hopital, Nice University Hospital, Nice